CLINICAL TRIAL: NCT06553924
Title: Single Dose Oral Bioequivalence Study of Macitentan and Tadalafil Film-coated Tablets 10 mg/40 mg and 'PrOpsynvi®' Macitentan and Tadalafil Film-coated Tablets 10 mg/40 mg in Healthy Adult Male Subjects Under Fasting Conditions
Brief Title: Macitentan and Tadalafil Film-coated Tablets 10 mg/40 mg and 'PrOpsynvi®' Macitentan and Tadalafil Film-coated Tablets 10 mg/40 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B03346
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: PAH
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macitentan and Tadalafil (Experimental): Macitentan and Tadalafil film-coated tablets 10 mg/40 mg
  Interventions: Drug: Macitentan and Tadalafil film-coated tablets; Drug: PrOpsynvi® macitentan and tadalafil film-coated tablets
- PrOpsynvi® film-coated tablets (Active Comparator): PrOpsynvi® macitentan and tadalafil film-coated tablets 10 mg/40 mg
  Interventions: Drug: Macitentan and Tadalafil film-coated tablets; Drug: PrOpsynvi® macitentan and tadalafil film-coated tablets

INTERVENTIONS:
Drug: Macitentan and Tadalafil film-coated tablets — 1 tablet of Macitentan and Tadalafil film-coated tablets 10 mg/40 mg
Drug: PrOpsynvi® macitentan and tadalafil film-coated tablets — 1 tablet of Macitentan and Tadalafil film-coated tablets 10 mg/40 mg

SUMMARY:
Single dose oral bioequivalence study of Macitentan and Tadalafil film-coated tablets 10 mg/40 mg and 'PrOpsynvi®' Macitentan and Tadalafil film-coated tablets 10 mg/40 mg in healthy adult male subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must fulfill all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified.

1) Age: 18 to 55 years old, both inclusive. 2) Gender: Male. 3) BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5). 4) Non-smokers and non-tobacco users (i.e. having no past history of smoking and tobacco consuming for at least one year prior to study).

5) Able to communicate effectively with study personnel. 6) Willing to provide written informed consent to participate in the study. 7) All volunteers must be judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which will include:

1. A physical examination (clinical examination) with no clinically significant finding.
2. Results within normal limits or clinically non-significant for the following tests: Hematology Hemoglobin Total RBC count Total WBC count Platelet count

   Differential leukocyte count:

   Neutrophils Lymphocytes Eosinophils Monocytes Basophils Blood indices: HCT Biochemistry BUN, Serum creatinine, Random glucose, SGPT & SGOT Alkaline phosphatase Uric acid Serum bilirubin Serum total protein: Total proteins, Albumin Serum electrolytes: Serum sodium, serum chloride, serum potassium, serum phosphorous, serum calcium Urinalysis Color, quantity, specific gravity, odour, appearance, reaction, albumin, bilirubin, ketone bodies, sugar, urobilinogen and microscopical examination (performed based on clinical judgment) Immunological Tests HIV-I & II, HbsAg ,Anti HCV
   * Additional tests and/or examinations (apart from mentioned in protocol) may be performed, if necessary, based on principal investigator discretion.
   * All results will be assessed against the current laboratory normal ranges at the time of testing and a copy of the normal ranges used will be included in the study documentation.

   EXCLUSION CRITERIA

   Volunteers must not be enrolled in the study if they meet any one of the following criteria:

   1) History of allergic responses to Macitentan, Tadalafil or other related drugs, or any of its formulation ingredients.

   Have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording].

   3) Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.

   4) History or presence of bronchial asthma. 5) Use of any hormone replacement therapy within 3 months prior to the first dose of study medication.

   6) Use of any depot injection or implant of any drug within 3 months prior to the first dose of study medication.

   7) Use of CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://drug interactions.medicine.iu.edu/MainTable.aspx). 8) History or evidence of drug dependence or of alcoholism or of moderate alcohol use.

   9) History of difficulty with donating blood or difficulty in accessibility of veins.

   10) A positive hepatitis screen (includes subtypes B & C). 11) A positive test result for HIV antibody. 12) Volunteers who have received an investigational drug within 90 days prior to the first dose of study medication.

   13) Volunteers who have donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever is greater.

   14) History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.

   15) Intolerance to venipuncture 16) Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.

   17) Institutionalized volunteers. 18) Use of any prescribed medications [Including guanylate cyclase stimulators, such as riociguat and potent CYP3A4 inhibitors (e.g. ritonavir, saquinavir, ketoconazole, itraconazole, and erythromycin)] within 14 days prior to the first dose of study medication.

   19) Use of any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.

   20) Use of grapefruit and grapefruit containing products within 7 days prior to the first döşe of study medication.

   Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeinecontaining sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products, dietary items that have effect on P450 enzymes (e.g. pomegranate, star fruit, seville oranges) & PGP (P-Glycoprotein) efflux pump (e.g. St. John's wort) within 48 hours prior to the first dose of study medication.

   22) Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.

   23) Use of any form of organic nitrate. 24) History of myocardial infarction, unstable angina or angina, heart failure, uncontrolled arrhythmias, hypotension, uncontrolled hypertension or stroke.

   25) Presence of anatomical deformation of the penis (such as angulation, cavernosal fibrosis, or Peyronie's disease).

   26) History or presence of benign prostatic hyperplasia. 27) History of vision loss or optic neuropathy. 28) Volunteer having Hemoglobin value lower than the lower limit of normal range during screening.

   29) SGPT, SGOT and alkaline phosphatase values 1.1 times higher than the upper limit of normal range during screening.

   30) Serum bilirubin value higher than the upper limit of normal range during screening.

   31) History of heart failure, pulmonary edema, fluid retention/peripheral edema, or chronic liver disease.

   32) History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 72 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00 - 125.00% for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time t (AUC0-t) | 72 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00 - 125.00% for each of the Ln-transformed data AUC0-t

SECONDARY OUTCOMES:
AUC from time 0 to infinity (AUCt-∞) | 72 hours
  Descriptive Statistics
Time to reach maximum concentration Cmax (Tmax) | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No